CLINICAL TRIAL: NCT06522256
Title: Identification of Molecular Signatures of High-risk Oncogenic HPV and Study of Their Associations With the Presence of High-grade Lesions and/or Anal Cancer 10 Years After Inclusion in the ANRS IPERGAY Trial
Acronym: HPVsign
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: INSERM SC10-US19 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS0251s-HPVSign
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: HPV Infection; Anal Cancer
Keywords: HSIL
MeSH Terms: conditions — Papillomavirus Infections; Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Transversal, non-comparative, multicenter study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-resolution anoscopy (Other)
  Interventions: Procedure: High-resolution anoscopy

INTERVENTIONS:
Procedure: High-resolution anoscopy — The study includes 2 visits:
  * a medical consultation for inclusion
  * a proctology consultation including the performance of an AHR associated or not with biopsy sampling

SUMMARY:
HPVsign is a cross-sectional, non-comparative, multicenter study involving all participants included in the HPV substudy of the ANRS IPERGAY trial. The study proposes to evaluate the cumulative incidence of high-grade lesions and/or anal cancers using high-resolution anoscopy (HRA) during the HPVsign study and/or diagnosed since the end of participation in the ANRS IPERGAY trial.

DETAILED DESCRIPTION:
The study aims to enrol 80 to 100 participants in French clinical centres. All the participants have participated to the IPERGAY HPV substudy.

The study proposes to evaluate the cumulative incidence of high-grade lesions and/or anal cancers using high-resolution anoscopy (HRA) during the HPVsign study and/or diagnosed since the end of participation in the ANRS IPERGAY trial.

Also, the study proposes to:

* study the association between the presence of HSIL and/or anal cancer and HPV molecular signatures during participation in the ANRS IPERGAY trial and 10 years after.
* study the evolution of HPV molecular signatures from participation in the ANRS IPERGAY to current study
* compare HRA results with anal cytology results
* compare the results of anal cytology concomitant with HRA with those obtained during participation in the ANRS IPERGAY trial.
* study factors associated with the presence of HSIL and/or anal cancer.
* compare the presence of different HPV virus types in the oropharynx concomitant with HRA and during participation in the ANRS IPERGAY trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the ANRS IPERGAY clinical trial who was included in the initial HPV sub-study;
* Informed and written signed consent
* Participant with regular health insurance

Exclusion Criteria:

* Participant under guardianship or curatorship
* Participant with free State medical assistance
* Participant who disagrees with the use of data collected as part of their participation in the ANRS IPERGAY trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
High-Grade Squamous Intraepithelial Lesion (HSIL) and/or anal cancers diagnosed by an high-resolution anoscopy (HRA) | Within the 10 years prior to HPV sign study participation, or at the study proctological examination in the study.

SECONDARY OUTCOMES:
HPV molecular signatures obtained using the Capture-HPV technique: HPV mutations, integration into the human genome | at the time of the ANRS IPERGAY-HPV sub-study, and 10 years later, in the HPVsign study.
Nature of abnormalities on High resolution anoscopy (HRA): condylomas, lesions. | 10 years after participation in the ANRS IPERGAY trial
  Lesions and condylomas are described as follows: location and type.
Nature of abnormalities on anal cytology: lesions location, lesions type, lesions grade. | at the time of the ANRS IPERGAY-HPV sub-study, and 10 years later, in the HPVsign study.
Nature of abnormalities on anal histology of lesions: location, type, grade | 10 years after participation in the ANRS IPERGAY trial
Presence of different HPV virus types in the oropharynx | at the time of the ANRS IPERGAY-HPV sub-study, and 10 years later, in the HPVsign study.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lascoux-Combe, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; David Veyer, Pharm D,PhD, Study Director — Hôpital Européen Georges-Pompidou
Locations (3):
- France (3):
  - Hôpital de la Croix Rousse - SMIT, Lyon
  - Hôpital Saint-Louis - SMIT, Paris
  - Hôpital Tenon - SMIT, Paris